CLINICAL TRIAL: NCT03526965
Title: Yoga Chikitsa for Neck Pain Caused by Cervical Spondylosis: a Randomized Controlled Pilot Trial
Brief Title: Yoga Chikitsa for Neck Pain Caused by Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/10124
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Chikitsa (Experimental): YC group were given traditional combination of yoga therapy including loosening movements, physical postures, breathing, relaxation and yoga counselling.
  Interventions: Other: Yoga Chikitsa; Drug: Usual care
- Usual Care (Active Comparator): Usual care were given exercise moves of necks, pain medications prescribed by physicians.
  Interventions: Drug: Usual care

INTERVENTIONS:
Other: Yoga Chikitsa — Intervention consisted of combination of static movements, yoga style exercise, yoga postures, breathing practices, relaxation and yoga counselling.
  Other Names: Yoga therapy
  Arms: Yoga Chikitsa
Drug: Usual care — Intervention included pain medications and exercise movements for neck.

SUMMARY:
Neck Pain caused by Cervical spondylosis (CS) is one of the most common health complaints. Despite its frequency as clinical problem worldwide, there are few evidence-based studies that document efficacy of therapies for neck pain. The aim of this study was to evaluate the effects of Yoga chikitsa (Yoga therapy) on pain and quality of life (QOL) in CS patients compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CS and confirmed by cervical radiographic examination
* Neck pain with CS
* Ready to Consent

Exclusion Criteria:

* Pregnancy
* Duration of neck pain < 6 months
* Comorbid systematic condition (Diabetes, Cardiovascular)
* History of cervical surgery, cervical injury, or disease of bones or joints.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Neck Pain | Change from baseline to 6 weeks
  Pain assessed by Northwick Park Neck Pain Questionnaire (NPQ)

SECONDARY OUTCOMES:
Quality of life | Change from baseline to 6 weeks
  Quality of life assessed by SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services; Manoj Swami, Principal Investigator — NMP Medical Research Institute
Locations (1):
- Pain Clinic, NMP Medical Research Institute, Jaipur, Rajasthan, India